CLINICAL TRIAL: NCT00541814
Title: Calcineurin Inhibitor Minimisation in Renal Transplant Recipients With Stable Allograft Function: A Prospective Randomised Controlled Trial
Brief Title: Calcineurin Inhibitor Minimisation in Renal Transplant Recipients With Stable Allograft Function
Acronym: CNIM-SRT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Birmingham (Other)
Collaborators: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RRK3367; ISRCTN No. 60081949
Record Dates: First submitted 2007-10-09; First posted 2007-10-10 (Estimated); Last update posted 2008-09-08 (Estimated); Status verified 2008-09

CONDITIONS: Chronic Allograft Nephropathy
Keywords: Renal Transplantation; Calcineurin Inhibitor; Cyclosporine; Withdrawal; Minimisation
MeSH Terms: interventions — Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): CNI [Cyclosporine] minimisation Group. Conversion from azathioprine to Myfortic followed by a three month period of cyclosporine weaning to target blood level of 50-100 ng/ml.
  Interventions: Drug: Cyclosporine
- 2 (Experimental): CNI [Cyclosporine] withdrawal Group. Conversion from azathioprine to Myfortic followed by a three month period of cyclosporine weaning to the point of withdrawal.
  Interventions: Drug: Cyclosporine

INTERVENTIONS:
Drug: Cyclosporine — Target drug level 50-100 ng/ml or cyclosporine withdrawal
  Other Names: Neoral

SUMMARY:
The purpose of this trial is to ascertain whether the withdrawal of calcineurin inhibitors (CNI) will lead to less kidney transplant damage when compared with minimisation. The investigators will assess this by comparing the degree of damage on kidney biopsies taken before and after minimisation/withdrawal of CNI.

DETAILED DESCRIPTION:
Renal transplantation is the most effective form of treatment for end-stage renal failure. It doubles long-term survival and has major socioeconomic and health benefits compared to patients who remain on dialysis. Graft survival in the UK is 90% at one year and greater than 75% at 5 years [UKTransplant, 2004], with better survival of grafts from living donors compared with deceased. However, by 15 years post-transplantation, over 50% of recipients who are still alive have returned to dialysis. Indeed, premature allograft failure is now one of the leading causes of end stage renal disease. As short-term outcomes of renal transplantation continue to improve, increasing attention is being paid to this late attrition of renal allografts.

It is recognised that calcineurin inhibitor (CNI) nephrotoxicity is a major factor in late renal allograft failure and dysfunction. In fact, withdrawal of CNI from patients with deteriorating graft function may improve graft function. However, there is abundant evidence that histological renal allograft damage may progress even in the absence of changes in renal function - i.e. declining renal function is a late marker of renal damage, and therefore institution of therapies (including CNI minimisation) to slow this process may be "too little, too late".

CNI minimisation may be optimised by three major routes. Firstly, by minimising the CNI beyond 12 months post transplantation when the risk of acute rejection is at its greatest. Secondly, by performing a renal biopsy in patients prior to CNI minimisation and avoiding CNI minimisation in patients with inflammation on the biopsy. Finally, converting azathioprine to mycophenolate prior to CNI minimisation should have a renoprotective effect.

The type of CNI we will investigate is cyclosporine.

Patients who fulfill the study entry criteria will require a renal allograft biopsy prior to randomisation to exclude acute rejection, recurrent disease or de novo glomerulonephritis. Those patients with an acceptable biopsy will proceed to randomisation on a 1:1 basis into 2 groups:

Group 1: CNI [Cyclosporine] minimisation; Group 2: CNI [Cyclosporine] withdrawal.

At this point participants will undergo assessment of the primary and secondary outcome measures. The treatment period comprises three stages:

Firstly, a 2 week period during which the patient will be stabilised on mycophenolate sodium 720mg twice daily (in place of azathioprine);

Secondly, a 3 month period during which the CNI [Cyclosporine} will be either targeted to a specified low blood level of 50-100ng/ml, or withdrawn completely (depending on randomisation);

Thirdly, a 12 month maintenance period on the new immunosuppression regimen.

During the first two stages, patients will be reviewed every 2 weeks. This 2-weekly follow-up will continue for the first two months of the third stage of the study, and then visits will be reduced to monthly. At these visits routine blood and urine analysis will be performed as per routine clinical practice.

At the end of the third stage of the study (i.e. 16 months after randomisation) the participants will undergo the second assessment of the primary and secondary outcome measures. This will signify study end for the individual study participant.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be an adult recipient of a first kidney transplant
* A functioning kidney allograft with estimated (e)GFR by MDRD > 30 ml/min/1.73 m2, and be between 1 and 5 years post transplantation
* Stable allograft function, as defined by no greater than 10% rise in serum creatinine in the preceding 6 months, on cyclosporine and azathioprine based immunosuppression
* Minimal proteinuria, evidenced as urine albumin: creatinine ratio < 50 mg/mmol

Exclusion Criteria:

* > = 18 years of age
* Pregnancy or suspicion of pregnancy confirmed by positive b-HCG pregnancy test
* Female patients unwilling to take effective contraception for study duration
* Untreated ureteric obstruction on ultrasound of allograft
* Recurrent urosepsis
* Severe systemic infection
* Untreated significant (> 50%) renal artery stenosis on magnetic resonance angiography performed prior to study
* History of acute allograft rejection
* History of myocardial infarction
* History of malignancy in previous 5 years (excluding non-melanomatous tumours limited to skin)
* Symptomatic ischaemic heart disease
* Hepatitis B surface antigen positive, Hepatitis C positive, or HIV positive
* Recipient of combined organ transplantation (e.g. pancreas/kidney; liver/kidney)
* Recipient of ABO-incompatible kidney
* Greater than 1 HLA mismatch at either the "B" or "DR" locus
* Peak HLA antibody Panel Reactivity (PRA) greater than 10%
* Recipient who underwent HLA desensitisation procedure prior to transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2007-10; Study Completion 2010-02 (Estimated)

PRIMARY OUTCOMES:
To compare renal allograft markers of damage and evolving injury in biopsies immediately pre study and at the end of the study | 16 months

SECONDARY OUTCOMES:
To compare markers of kidney transplant function | 16 months
To compare markers of immune function | 16 months
Infection episodes | 16 months
To assess changes in independent cardiovascular risk factors | 16 months
Malignancy | 16 months
Patient Survival | 16 months

CONTACTS AND LOCATIONS:
Overall Officials: Richard Borrows, MRCP, Principal Investigator — University Hospital Birmingham NHS Foundation Trust
Locations (1):
- University Hospital Birmingham NHS Foundation Trust, Birmingham, West Midlands, United Kingdom

REFERENCES:
- See also: Sponsor website — http://www.uhb.nhs.uk